CLINICAL TRIAL: NCT07012148
Title: FORESITE (FOREcasting Seizures to Initiate ThErapy): Optimizing Management of Drug-Resistant Epilepsy Using Seizure Forecasts Via Subscalp EEG and Wearables
Brief Title: Optimizing Therapy in Epilepsy Using Seizure Forecasts Via EEG and Wearables
Acronym: FORESITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Benjamin H. Brinkmann, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23-005125; UG3NS123066-02 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy; Generalized Seizure; Drug Refractory Epilepsy
Keywords: complex partial seizure; UNEEG; seizure forecasting; Subscalp EEG
MeSH Terms: conditions — Epilepsies, Partial; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: All study participants will be implanted with a subscalp EEG system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- subscalp EEG (Experimental): All study subjects will be implanted with the UNEEG SubQ device.
  Interventions: Device: UNEEG SubQ device

INTERVENTIONS:
Device: UNEEG SubQ device — Subjects will be implanted with the UNEEG SubQ device in the neurosurgical operating suite under general anesthesia. Electrodes will be placed over the temporal lobe of the hemisphere established as the origin of seizures by previous EEG monitoring. Only one UNEEG device will be placed, and only the seizure onset hemisphere will be covered.

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of using seizure forecasts based on subscalp EEG.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must have epilepsy involving the temporal lobe and will have undergone video-EEG monitoring within the past 3 years, and will have met the following criteria:

* Focal epilepsy, including complex partial, and secondarily generalized seizures, including:

  * disabling seizure (i.e. involving loss of awareness, motor control, speech, or other essential functions) counts at least 2 per month on average over the preceding 3 months, established by verbal history or caregiver report.
  * For 3 months prior to enrollment, subject's AED dosages have been stable (less than a 25% change in dosage) and subject has had at least two seizures per month, on average, with a seizure-free interval not to exceed 60 days. Seizures must be separated by a minimum of four hours not to be considered part of a cluster. A cluster, for the purpose of this criterion, shall be considered a single seizure.
* With the exception of epilepsy, subject must be medically and neurologically stable.
* Age 18 to 75.
* Ability and willingness to provide informed consent and participate in the study protocol. Subject is able to interpret and to respond, in accordance with the study protocol, to the advisory indicators provided by the device.
* Subject has seizures that are distinct, stereotypical events that can be reliably counted by the subject or caregiver, and have a distinct EEG pattern that can be recorded using subscalp EEG over the frontotemporal head region, established by video-EEG monitoring.
* Subject can reasonably be expected to maintain a seizure diary alone or with the assistance of a competent individual.
* Subject is able to complete regular office visits and telephone appointments in accordance with the study protocol requirements.
* Subject's seizure focus, based upon clinical semiology, scalp EEG, intracranial electroencephalographic (iEEG) findings, and/or neuroimaging, demonstrate consistent involvement of the temporal lobe with their EEG seizure pattern.
* Subject speaks and reads English.
* Subject has no reason to anticipate requiring a magnetic resonance imaging (MRI) evaluation within the next two years.
* Subject has EEG documentation of ictal events consistent with his or her predominant current seizure type.
* Subject's anatomy will permit implantation of the UNEEG SubQ device in the opinion of the study's neurosurgeon.
* Female subjects have a negative pregnancy test, have no plans to become pregnant, and use effective contraception during the study.

Exclusion Criteria:

* For 3 months prior to enrollment, subject's AED dosages have not been stable (greater than 25% change in dosage), or subject has had more than 30 disabling seizures per month, on average, or more than 10 seizure days per month, on average.
* Subject needs to have magnetic resonance imaging during the study period.
* Subject has a substance abuse history (alcohol, prescription, or illicit medications) within the preceding two years.
* Subject participated in another drug or device trial within the preceding 30 days.
* Subject has been hospitalized for a psychiatric condition within the preceding two years or has had a history of psychosis within the preceding two years (excluding post-ictal psychosis).
* Subject is implanted with pacemaker, implantable cardiac defibrillator, cardiac management product, brain stimulator, or other medical device that would interfere with the UNEEG device. This includes, but is not limited to, direct brain neurostimulators, spinal cord stimulators, and cochlear implants. Vagus nerve stimulators are not expected to interfere with the subscalp EEG device and will be permitted, as long as stimulation parameters can be reasonably expected to remain stable (25% or less change in amplitude) throughout the study.
* Subject has experienced unprovoked status epilepticus.
* Subject has had therapeutic surgery to treat epilepsy that may interfere with electrode placement in the judgement of the neurosurgeon.
* Subject is on anticoagulants and is unable to discontinue them perisurgically, as required by the neurosurgeon or Investigator.
* Subject has significant platelet dysfunction from medical conditions or medications (including, particularly, aspirin or sodium valproate). If platelet dysfunction is suspected, subject can be enrolled only if a hematologist, the Investigator, and the neurosurgeon judge it to be advisable. Blood tests to evaluate platelet and bleeding disorder issues will be obtained prior to enrollment.
* Subject is otherwise ineligible for cranial surgery, or the Investigators identify other medical or psychosocial factors that would counter indicate participation in the study.
* Subject is pregnant or intends to become pregnant during the study period.
* Subject has a known diagnosis of psychogenic nonepileptic seizures (PNES)
* Female subject is pregnant or plans to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events | 12 months
  Number of device-related adverse events during the study period
Surgical and Device related adverse events | 12 months
  Following surgery adverse events related to surgery and the device will be assessed, including: pain/soreness at the surgical site up to 1 week after surgery, pain/soreness at the surgical site after more than 1 week after surgery, headache (nonsurgical), skin irritation at transceiver position, excess bleeding, and infection; additionally, skin erosion will be assessed, and lead migration and fracture will be assessed by x-ray, if there is any concern for this, at the time of study completion prior to explantation.

SECONDARY OUTCOMES:
Quality of Life Inventory | 12 months
  The Quality of Life Inventory in Epilepsy (QOLIE-31) contains seven multi-item scales across the domains of emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, and overall quality of life. Scoring of the QOLIE-31 requires the conversion of raw data to a scale of 0 to 100 for each sub-scale, with higher scores reflecting higher quality of life
  Timeframe: Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brinkmann, PhD, Principal Investigator — Mayo Clinic; Gregory A Worrell, MD, PhD, Principal Investigator — Mayo Clinic; Jamie J Van Gompel, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pal Attia T, Viana PF, Nasseri M, Duun-Henriksen J, Biondi A, Winston JS, P Martins I, Nurse ES, Dumpelmann M, Worrell GA, Schulze-Bonhage A, Freestone DR, Kjaer TW, Brinkmann BH, Richardson MP. Seizure forecasting using minimally invasive, ultra-long-term subcutaneous EEG: Generalizable cross-patient models. Epilepsia. 2023 Dec;64 Suppl 4(Suppl 4):S114-S123. doi: 10.1111/epi.17265. Epub 2022 May 4. PMID 35441703
- [Background] Viana PF, Pal Attia T, Nasseri M, Duun-Henriksen J, Biondi A, Winston JS, Pavao Martins I, Nurse ES, Dumpelmann M, Schulze-Bonhage A, Freestone DR, Kjaer TW, Richardson MP, Brinkmann BH. Seizure forecasting using minimally invasive, ultra-long-term subcutaneous electroencephalography: Individualized intrapatient models. Epilepsia. 2023 Dec;64 Suppl 4(Suppl 4):S124-S133. doi: 10.1111/epi.17252. Epub 2022 Apr 16. PMID 35395101
- [Background] Nasseri M, Stirling RE, Viana PF, Cui J, Nurse E, Karoly PJ, Kremen V, Dumpelmann M, Worrell GA, Freestone DR, Richardson MP, Brinkmann BH. Forecasting epileptic seizures with wearable devices: A hybrid short- and long-horizon pseudo-prospective approach. Epilepsia. 2025 Sep;66(9):3293-3308. doi: 10.1111/epi.18466. Epub 2025 May 24. PMID 40411751
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials